CLINICAL TRIAL: NCT01500863
Title: Endometrial Receptivity After GnRH Agonist Triggering From Final Oocyte Maturation
Brief Title: Endometrial Receptivity After GnRH Agonist Triggering
Acronym: ERAMAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MAD-AB-ERA-2011
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: endometrial receptivity; gene arrays; agonist triggering; Endometrial gene expression; OHSS
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Triptorelin Pamoate; Estradiol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- hCG (Active Comparator)
  Interventions: Drug: hCG
- Triptorelin 0.2mg s.c. (Experimental)
  Interventions: Drug: triptorelin
- 0.2mg triptorelin plus estradiol/progesterone (Experimental)
  Interventions: Drug: Triptorelin, estradiol valerate, micronized vaginal progesterone
- 0.2mg tripoterlin plus single bolus hCG 1500 IU (Experimental)
  Interventions: Drug: triptorelin, hCG
- 0.2mg tripoterlin plus multiple boluses hCG 500 IU (Experimental)
  Interventions: Drug: triptorelin, hCG
- 0.2mg tripoterlin plus multiple doses recLH (Experimental)
  Interventions: Drug: triptorelin, recombinant LH

INTERVENTIONS:
Drug: hCG — single shot of 6500 IU hCG s.c. at the time of triggering
  Arms: hCG
Drug: triptorelin — single shot of 0.2mg triptorelin s.c. at the time of triggering
  Arms: Triptorelin 0.2mg s.c.
Drug: Triptorelin, estradiol valerate, micronized vaginal progesterone — 4mg of estradiol valerate per os plus 400mg micronized vaginal progesterone daily starting the day after OPU
  Arms: 0.2mg triptorelin plus estradiol/progesterone
Drug: triptorelin, hCG — single shot of 1500 IU hCG s.c. the day of OPU plus 4mg of estradiol valerate per os plus 400mg micronized vaginal progesterone daily starting the day after OPU
  Arms: 0.2mg tripoterlin plus single bolus hCG 1500 IU
Drug: triptorelin, hCG — Multiple doses of 500 IU hCG (OPU, +4 and +7) and 4mg of estradiol valerate per os plus 400mg micronized vaginal progesterone daily starting the day after OPU
  Arms: 0.2mg tripoterlin plus multiple boluses hCG 500 IU
Drug: triptorelin, recombinant LH — 300 IU recombinant LH every 48h and 4mg of estradiol valerate per os plus 400mg micronized vaginal progesterone daily starting the day after OPU
  Arms: 0.2mg tripoterlin plus multiple doses recLH

SUMMARY:
Conventional luteal phase support after human chorionic gonadotrophin (hCG) triggering in women undergoing in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) provides adequate pregnancy rates and live birth rates, but Ovarian hyperstimulation syndrome (OHSS) still occurs in 1-3% of the patients. If gonadotropin-releasing hormone agonist (GnRHa) are used instead of hCG, OHSS does not occur, but clinical results are somehow diminished.

By testing different luteal support protocols on women undergoing GnRHa triggering, the investigators aim to find out which protocol resembles the most the gene expression profile observed after hCG triggering and conventional luteal phase support, in order to choose it as the most adequate in terms of endometrium receptivity and safety (OHSS incidence).

ELIGIBILITY:
Inclusion criteria :

* Healthy oocyte donor women
* Aged 18-35 years
* With a menstrual cycle length of 26-35 days
* Normal ultrasound scan of uterus and ovaries
* Normal basal hormones
* No contraindication for controlled ovarian stimulation (COS)
* Willing to participate in the study and providing written informed consent.

Exclusion Criteria:

* Subjects with current or previous history of an endocrine abnormality
* Subjects with an abnormal outcome of blood biochemistry or hematology
* Subjects with an abnormal cervical smear
* Subjects with a chronic disease
* Subjects with any relevant ovarian-, tubal- or uterine-pathology that could interfere with the COS treatment
* Pregnancy
* Subjects who had a previous history of ovarian hyperresponse or ovarian hyperstimulation syndrome (OHSS), polycystic ovary syndrome (PCOS) or a basal antral follicle count (AFC) of more than 20 on ultrasound (11 mm, both ovaries combined) .
* Previous low ovarian response to FSH or hMG treatment (i.e. cycle cancelled due to insufficient ovarian response or less than 6 oocytes obtained).
* A history of recurrent miscarriage,
* Smoking more than 10 cigarettes per day.
* Not willing to comply with study procedures

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
endometrial receptivity gene expression profile | participants will be followed for the duration of the cycle, an expected average of 4 weeks

SECONDARY OUTCOMES:
Incidence of moderate/severe OHSS in all different treatment group | participants will be followed for the duration of the cycle, an expected average of 4 weeks
  Mild OHSS Grade 1, abdominal distension and discomfort Grade 2, features of grade 1 plus nausea, vomiting and/or diarrhea; ovaries are enlarged from 5 to 12 cm Moderate OHSS Grade 3, features of mild OHSS plus ultrasonic evidence of ascites Severe OHSS Grade 4, features of moderate OHSS plus evidence of ascites and/or hydrothorax and breathing difficulties Grade 5, all of the above, plus change in the blood volume, increased blood viscosity due to hemoconcentration, coagulation abnormality, and diminished renal perfusion and function

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Bermejo, MD, Study Director — IVI Madrid
Locations (1):
- Instituto Valenciano de Infertilidad, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No